CLINICAL TRIAL: NCT03689504
Title: Evaluating a Family-based Nutrition and Garden Intervention in Rural Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuqu' Kawoq, Maya Health Alliance (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WK-2018-002
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Malnutrition; Dietary Modification
Keywords: Guatemala; indigenous; dietary diversity; chronic malnutrition; Maya; agriculture; behavior change; food insecurity
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): The standard of care is an intensive individualized home-based nutrition education program, together with a home food ration and micronutrient supplement, delivered by frontline workers for 6 months.
  Interventions: Dietary Supplement: Standard of care nutrition support; Behavioral: Home-based nutrition education
- Home Garden Intervention (Experimental): This arm adds an 8 month individualized home-based family garden intervention to the existing standard of care (home-based nutrition education)
  Interventions: Dietary Supplement: Standard of care nutrition support; Behavioral: Home-based nutrition education; Behavioral: Home-based family gardening

INTERVENTIONS:
Dietary Supplement: Standard of care nutrition support — Subjects will be provided with a standard food ration and with a multiple micronutrient powder (Chispitas) or lipid-based nutrient supplement (Nutributter)
Behavioral: Home-based nutrition education — Health promoters will use 24-hour dietary recall information to assess meal frequency and dietary diversity and then provide tailored nutrition coaching to parents.
Behavioral: Home-based family gardening — Health promoters will facilitate the building and maintenance of a family home garden using a square foot or container gardening method.
  Arms: Home Garden Intervention

SUMMARY:
This is a pilot quasi-experimental study to evaluate the impact of adding a family garden intervention to an existing wrap-around nutrition intervention for children with chronic malnutrition and their family. The existing nutrition intervention is provided by community health workers affiliated with Wuqu' Kawoq | Maya Health Alliance. A single community in rural Guatemala will participate in the intervention, with the goal to recruit approximately 70 families in the combined nutrition/garden intervention. A nearby community, also participating in the nutrition intervention, will serve as a nonrandom contemporaneous control.

Aims of the study include:

1. Evaluate the impact of the garden intervention on maternal and child dietary diversity, child growth and household food insecurity.
2. Use the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework to conduct a preliminary implementation analysis, to guide a future, well-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Children who are already scheduled to be enrolled in Maya Health Alliance's intensive home-based nutrition program (non-investigational, standard of care) who are 6-24 months of age at the time of enrollment with a height-for-age Z scores of <= -2.5
* At least one caregiver willing to provide written informed consent
* Caregiver of a child enrolled in the study (for caregiver/head of household outcomes), including women who may be pregnant
* Planned residence in the study area for the next 18 months

Exclusion Criteria:

* Children with acute malnutrition (weight for length Z scores of <= -2.0)
* Children with a severe medical illness that affects growth (e.g., heart disease, kidney disease, genetic condition) as determined by a Maya Health Alliance staff physician.
* Caregivers with cognitive impairments that prevent them from being able to provide informed consent

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rohloff, MD PhD, Principal Investigator — Wuqu' Kawoq; Beth Jimenez, RDN PhD, Principal Investigator — University of New Mexico; Andrea Guzman, RDN, Study Director — Wuqu' Kawoq
Locations (1):
- Wuqu' Kawoq, Tecpán Guatemala, Departamento de Chimaltenango, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified demographic, clinical, and outcomes will be made available on a public data repository after completion of primary analysis and at the time of publication of results manuscripts.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Supporting data will be shared indefinitely on public data repositories at the time of manuscript publication.
Access Criteria: Publicly available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Home Garden Intervention
Started | 70 | 70
Completed | 65 | 70
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Home Garden Intervention | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 376 [265 to 524] | 343 [259 to 471] | 353 [262 to 502]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 38 | 41 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: data missing
  Participants
    Maya ethnicity/language preference: number analyzed (Participants) | 69 | 70 | 139
    Maya ethnicity/language preference | 65 | 68 | 133
Region of Enrollment [Number; unit: participants]
  Guatemala | 70 | 70 | 140
Length for age Z score [Median (Inter-Quartile Range); unit: Z score] — These are z-scores calculated against the World Health Organization pediatric growth reference population (https://www.who.int/tools/child-growth-standards/standards)
  Z score | -3.05 [-3.57 to -2.68] | -3.20 [-3.7 to -2.68] | -3.15 [-3.64 to -2.68]
Weight for age Z score [Median (Inter-Quartile Range); unit: Z score] — These are z-scores calculated against the World Health Organization pediatric growth reference population (https://www.who.int/tools/child-growth-standards/standards)
  Z score | -1.55 [-2.07 to -1.25] | -1.58 [-2.23 to -1.07] | -1.56 [-2.14 to -1.07]
Weight for length Z score [Median (Inter-Quartile Range); unit: Z score] — These are z-scores calculated against the World Health Organization pediatric growth reference population (https://www.who.int/tools/child-growth-standards/standards)
  Z score | 0.18 [-0.30 to 0.75] | 0.32 [-0.18 to 0.86] | 0.3 [-0.28 to 0.79]
Minimum acceptable diet [Count of Participants; unit: Participants] — This is a composite diet quality measure developed by the World Health Organization in the technical manual Infant and Young Child Feeding Indicators. It references achieving both minimum recommended food group consumption and solid meal consumption within a 24 hour recall period, with adjustments for age and breastfeeding status. Full details: https://www.who.int/publications/i/item/9789240018389
  Participants | 34 | 48 | 82

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Food Groups Consumed Per Day at 6 Months - Child
Description: Calculated from the World Health Organization Infant and Young Child Feeding Indicators 24 hour diet recall tool
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: food groups
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 64
food groups | 0.6 (1.84) | 1.29 (1.59)

2. Primary Outcome: Change From Baseline in Mean Number of Solid Meals Consumed Per Day at 6 Months - Child
Description: Calculated from the World Health Organization Infant and Young Child Feeding Indicators 24 hour diet recall tool
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: solid meals
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 70
solid meals | 0.81 (1.61) | 1.11 (1.45)

3. Primary Outcome: Change From Baseline in Raw Household Food Insecurity Score at 6 Months
Description: Standardized food insecurity score, using the Food and Agriculture Organization's Global Food Insecurity Experience Scale (possible score range 0-8), higher scores indicate more food insecurity
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 64
score on a scale | -0.55 (1.86) | -0.84 (2.1)

4. Primary Outcome: Change From Baseline in Mean Number of Food Groups Consumed Per Day at 6 Months - Female Head of Household
Description: Calculated from the Food and Agriculture Organization's Minimum Dietary Diversity for Women dietary recall
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: food groups
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 64
food groups | -0.01 (1.88) | 0.42 (1.75)

5. Secondary Outcome: Change in Height/Length for Age Z Score From Baseline to 6 Months
Description: These are differences from 0 to 6 months (baseline to 6 months of intervention) z-scores calculated against the World Health Organization pediatric growth reference population (https://www.who.int/tools/child-growth-standards/standards)
Time Frame: 0 months (baseline), 6 months
Measure: Mean (Standard Deviation); unit: change in Z score
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 64
change in Z score | -0.21 (0.49) | -0.07 (0.51)

6. Secondary Outcome: Change in Weight for Age Z Score From Baseline to 6 Months
Description: as for outcome 5
Time Frame: 0 months (Baseline), 6 months
Measure: Mean (Standard Deviation); unit: Change in Z score
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 64
Change in Z score | -0.22 (0.39) | -0.12 (0.29)

7. Secondary Outcome: Change in Weight for Height/Length Z Score From Baseline to 6 Months
Description: as for outcome 5
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Change in Z score
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 64
Change in Z score | -0.38 (0.64) | -0.24 (0.54)

8. Secondary Outcome: Mean Change in Household Crop Species From Baseline to 6 Months Diversity Score
Description: Raw count of total crop species cultivated in the home
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: crop species
Arm/Group | Standard of Care | Home Garden Intervention
Number analyzed (Participants) | 70 | 64
crop species | -1.1 (4.15) | 4.62 (4.66)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard of Care | Home Garden Intervention
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03689504/Prot_SAP_000.pdf